CLINICAL TRIAL: NCT01752972
Title: Effect of Spirulina on the Levels of Zinc, Vitamin E and Linoleic Acid in the Palm Skin Extracts of People With Prolonged Exposure to Arsenic
Brief Title: Effect of Spirulina on Zinc, Vitamin E and Linoleic Acid Levels in Palm Skin Following Chronic Exposure to Arsenic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Mir Misbahuddin, Prof. and Chairman, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BSMMU-006-CT
Record Dates: First submitted 2012-12-17; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Arsenical Keratosis
Keywords: Arsenic; Keratosis; Linoleic acid; Palm; Spirulina; Vitamin E; Zinc
MeSH Terms: conditions — Keratosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Palmer arsenical keratosis (Experimental): Spirulina 10 g/day orally for 12 weeks
  Interventions: Dietary Supplement: Spirulina
- Arsenic exposed controls (Active Comparator): Spirulina 10 g/day orally for 12 weeks
  Interventions: Dietary Supplement: Spirulina
- Heathy volunteers (Active Comparator): Spirulina 10 g/day orally for 12 weeks
  Interventions: Dietary Supplement: Spirulina

INTERVENTIONS:
Dietary Supplement: Spirulina — 10 g/day orally for 12 weeks

SUMMARY:
Patients of arsenical keratosis may be treated with spirulina. Is this improvement related to the levels of zinc, vitamin E and linoleic acid at the site of the keratosis (palm)? To understand this, patients of palmer arsenical keratosis (n=10), arsenic exposed controls (n=10) and healthy volunteers (n=10) will be treated with spirulina powder 10 g/day orally for 12 weeks. Skin extracts will be collected both before and after supplementation from the palm and dorsum for estimation of zinc, vitamin E and linoleic acid levels.

DETAILED DESCRIPTION:
Patients of arsenical keratosis remain untreated due to unavailability of effective drug. To find out an effective drug, the pathogenesis of keratosis should be understood. Spirulina is one of the dietary supplements, that improves the symptoms of keratosis. Is this improvement related to the levels of zinc, vitamin E and linoleic acid at the site of the keratosis (palm)? Ten patients of moderate palmer arsenical keratosis will be treated with spirulina powder 10 g/day orally for 12 weeks. Skin extracts will be collected both before and after supplementation from the palm and dorsum using a mixture of chloroform and ethanol. Zinc, vitamin E and linoleic acid levels will be estimated from the extracts. Similar protocol of spirulina administration and the collection of skin extracts will be done in arsenic exposed controls (n=10) and healthy volunteers (n=10).

ELIGIBILITY:
Inclusion Criteria (Patients):

* moderate palmer keratosis
* drink arsenic contaminated water (>50 µg/L) for at least 6 months
* voluntarily agree to participate

Inclusion Criteria (Arsenic exposed controls):

* no symptoms of keratosis
* family member of the patient
* drink arsenic contaminated water (>50 µg/L) for at least 6 months
* voluntarily agree to participate

Inclusion Criteria (Healthy volunteers):

* no symptoms of keratosis
* drink arsenic safe water (<50 µg/L)
* voluntarily agree to participate

Exclusion Criteria:

* pregnancy
* lactation
* chronic diseases: diabetes mellitus, rheumatoid arthritis, tuberculosis
* arsenicosis patients under treatment in the previous 3 months

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in vitamin E levels in skin palm extract following supplementation with spirulina | 0 week (baseline), 12 weeks (end)

SECONDARY OUTCOMES:
Change in zinc levels in skin palm extract following supplementation with spirulina | 0 week (baseline), 12 weeks (end)
Change in linoleic acid levels in skin palm extract following supplementation with spirulina | 0 week (baseline), 12 weeks (end)

CONTACTS AND LOCATIONS:
Overall Officials: Mir Misbahuddin, MBBS, PhD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh